CLINICAL TRIAL: NCT03337490
Title: A Randomized, Multi-Center, Double-blind, Placebo Controlled, Parallel Group Trial to Evaluate Efficacy and Safety of Mayne Pharma's Ivermectin 0.5% Lotion Compared to Sklice® Ivermectin 0.5% Lotion in the Treatment of Head Lice
Brief Title: A Clinical Endpoint Bioequivalence Study to Assess Efficacy and Safety of Ivermectin 0.5% Lotion in the Treatment of Head Lice
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayne Pharma International Pty Ltd (Industry)
Collaborators: bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAP-7189
Record Dates: First submitted 2017-10-30; First posted 2017-11-09 (Actual); Results first posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Head Lice
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ivermectin 0.5% Lotion (Experimental): Ivermectin 0.5% lotion, topical, 117g, single dose
  Interventions: Drug: Ivermectin 0.5% Topical Application Lotion
- Ivermectin 0.5% Lotion [SKLICE] (Active Comparator): Sklice 0.5% Lotion, topical, 117g, single dose
  Interventions: Drug: Ivermectin 0.5% Topical Application Lotion [SKLICE]
- Placebo 0% Lotion (Placebo Comparator): 0% lotion, 117g, single dose
  Interventions: Drug: Placebo 0% Lotion

INTERVENTIONS:
Drug: Ivermectin 0.5% Topical Application Lotion — Subjects on Test Product will receive a single dose, 117g, during the study to be applied at baseline.
  Arms: Ivermectin 0.5% Lotion
Drug: Ivermectin 0.5% Topical Application Lotion [SKLICE] — Subjects on Reference Product will receive a single dose, 117g, during the study to be applied at baseline.
  Arms: Ivermectin 0.5% Lotion [SKLICE]
Drug: Placebo 0% Lotion — Subjects on Placebo will receive a single dose, 117g, during the study to be applied at baseline.
  Arms: Placebo 0% Lotion

SUMMARY:
This is a phase 3 randomized, multi-center, double-blind, placebo controlled, parallel group design study.

DETAILED DESCRIPTION:
This study is comprised of two phases: screening and treatment. The screening period is 24 hours, followed by the treatment phase of 15 ± 3 days. During the treatment phase, subjects will be randomized to either test, reference of placebo treatments (3:3:1) in a double-blind manner in an outpatient setting. Once eligibility is confirmed, randomization will occur at visit 2 (baseline, Day 1) i.e. initiation of treatment phase. The treatment phase will be 15 ± 3 days in duration wherein subject will receive treatment with investigational product (either test, reference or placebo) on Day 1 or baseline (visit 2). Efficacy will be evaluated at Day 15. Safety and tolerability will be evaluated based upon AEs and patient self-assessments and self-assessments collected during follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have an active head lice infestation defined as: At least 3 live lice (adults and/or nymphs) present on the scalp and/or hair, as determined by a trained evaluator. The index subject must be the youngest family member, through the age of 18, presenting with an active head lice infestation.
2. Household members that have an active head lice infestation defined as: At least 1 live louse (adult and/or nymph) present on the scalp and/or hair, as determined by a trained evaluator (with the exception of the male head of household who may self-assess as being lice free) will receive the Standard of Care with an over-the-counter head lice treatment product. Up to 3 infested household members may receive treatment, if more than 3 household members are infested, the entire household will be excluded from the study.
3. Subject is male or female.
4. Index subject is at least 6 months through 18 years of age at time of enrollment.
5. Subject is in good general health based on medical history.
6. Each subject must have an appropriately signed Informed Consent agreement. A caregiver must sign an Informed Consent agreement for children not old enough to do so. Children ages 6-17 years of age will be administered a child's Assent Form.
7. The caregiver of a subject must be willing to allow all household members to be screened for head lice. If other household members are found to have an active head lice infestation, they must be willing and able to participate in receiving the Standard of Care. No more than one working male per household may be excluded from evaluation if he is assessed as being lice free by himself or the caregiver and cannot come in due to his work schedule. If this individual may have lice, he must come to the test facility; otherwise the entire household will be excluded from study participation.
8. Subject and/or their caregiver must be physically able and willing to apply the test product according to established treatment methods.
9. Subject agrees not to use any other form of lice treatments (commercial, community-anecdotal, or mechanical/manual) while participating in the study.
10. Following application and rinsing of the test product, subject agrees not to shampoo, wash, or rinse their hair or scalp until the 24-hour post-treatment evaluation has been completed.
11. Subject agrees to not cut or chemically treat their hair while participating in the study.
12. Subject agrees to follow all study instructions, including attending all follow-up appointments.
13. Female index subjects of childbearing potential must be willing to have a urine pregnancy test prior to inclusion in this study.
14. In the event of a subject judged to be incapable of self-treating, the household must have a caregiver willing to apply the treatment at home.

Exclusion Criteria:

1. Index subjects with greater than 3 household members with at least 1 live louse (adult and/or nymph) present on the scalp and/or hair, as determined by a trained evaluator will be automatically excluded from the trial.
2. Youngest household member is over 18 years of age.
3. History of irritation or sensitivity to ivermectin or the lotion components, pediculicides or hair care products.
4. Presentation at the treatment site with visible skin/scalp condition(s) that are not attributable to head lice infestation, such as an erythema score that is >2, blisters, vesicles which, in the opinion of the investigative personnel or medical monitor, will interfere with safety and/or efficacy evaluations.
5. Presentation at the treatment site with eczema or atopic dermatitis.
6. Treatment for head lice (Over the counter [OTC], home remedy and/or Prescription) in the last 15 days.
7. Any condition or illness that, in the opinion of the investigator, may compromise the objective of the protocol.
8. Is receiving any other treatment which, in the opinion of the investigator or medical monitor, may interfere with the study results.
9. Females (including caregivers who come in contact with the investigational product) who are pregnant, nursing or planning a pregnancy which could include index subjects. If a household has a pregnant female who has an active case of lice, the entire household is excluded from participation. If this pregnant household member does not have an active infestation, this individual must NOT be the caregiver (one who provides treatment to other household members).
10. Index subject of child-bearing potential, and unwilling to use an adequate method of contraception for the duration of the study. Adequate methods of contraception include: abstinence, vasectomized partner, oral birth control pills, birth control injections or patches, Intra uterine devices, condoms with a spermicidal jelly or a diaphragm with spermicidal jelly, surgical sterilization. Index subjects and/or their caregivers will be considered non-child-bearing if the following has occurred: full hysterectomy or bilateral oophorectomy is considered surgically sterile. Tubal ligation is not considered equivalent to female sterilization.
11. Participation in a previous investigational drug study within the past 30 days.
12. Does not understand the requirements for study participation and/or may likely exhibit poor compliance, in the opinion of the investigator.
13. Does not have a known household affiliation with their household members (i.e., do not stay in one household consistently, sleeping at one place several nights and then at another place or location). Household is defined as living in a shared area or space (for example the same house or apartment unit).

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 296 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Site 105, Dinuba, California
  - Site 104, Miami, Florida
  - Site 101, Plantation, Florida
  - Site 102, West Palm Beach, Florida
  - Site 106, Nashville, Tennessee
  - Site 103, Richland, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ivermectin 0.5% Lotion | Ivermectin 0.5% Lotion [SKLICE] | Placebo 0% Lotion
Started | 128 | 126 | 42
Completed | 117 | 112 | 7
Not Completed | 11 | 14 | 35
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lack of Efficacy | 10 | 12 | 35
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 1 subject in the Ivermectin 0.5% Lotion [SKLICE] arm was not part of the mITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivermectin 0.5% Lotion | Ivermectin 0.5% Lotion [SKLICE] | Placebo 0% Lotion | Total
Number analyzed (Participants) | 128 | 125 | 42 | 295
Age, Customized [Count of Participants; unit: Participants]
  1 Month-2 Years | 2 | 11 | 3 | 16
  2-12 Years | 89 | 73 | 27 | 189
  12-16 Years | 22 | 22 | 6 | 50
  =>16 Years | 15 | 19 | 6 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 91 | 29 | 208
  Male | 40 | 34 | 13 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska native | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 1 | 6
  White | 118 | 115 | 39 | 272
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Other/missing | 6 | 8 | 2 | 16
  Hispanic or Latino | 102 | 105 | 35 | 242
  Not Hispanic or Latino | 11 | 9 | 3 | 23
  Missing | 15 | 11 | 4 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 128 | 125 | 42 | 295
Head Lice Visual Assessment [Count of Participants; unit: Participants] | 128 | 125 | 42 | 295

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Index Subjects Who Are Lice Free at Day 15
Description: The primary endpoint is the proportion of index subjects who are lice free at Day 15
Time Frame: 15 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Ivermectin 0.5% Lotion | Ivermectin 0.5% Lotion [SKLICE] | Placebo 0% Lotion
Number analyzed (Participants) | 115 | 111 | 40
Participants | 106 | 98 | 7

2. Secondary Outcome: The Number of All Index Subjects Who Are Lice-free at Day 2
Description: The secondary endpoint includes the number of all index subjects who are lice-free at Day 2
Time Frame: 2 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Ivermectin 0.5% Lotion | Ivermectin 0.5% Lotion [SKLICE] | Placebo 0% Lotion
Number analyzed (Participants) | 115 | 111 | 40
Participants | 112 | 109 | 10

ADVERSE EVENTS:
Time Frame: 2.5 months from first subject first visit.
Description: No deaths or serious adverse events occurred during the duration of this study.
Arm/Group | Ivermectin 0.5% Lotion | Ivermectin 0.5% Lotion [SKLICE] | Placebo 0% Lotion
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/125 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/125 | 0/42
Other Adverse Events (participants affected / at risk) | 0/128 | 3/125 | 2/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivermectin 0.5% Lotion (N=128) | Ivermectin 0.5% Lotion [SKLICE] (N=125) | Placebo 0% Lotion (N=42)
Pyrexia (General disorders) | 0 | 0 | 1
Upper Resporitory Tract Infection (General disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT03337490/SAP_000.pdf
  • Study Protocol (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT03337490/Prot_001.pdf